CLINICAL TRIAL: NCT04142541
Title: Protection Against Emboli During Carotid Artery Stenting Using a 3-in-1delivery System Comprised of a Post-dilation Balloon, Integrated Embolic Filter, and a Novel Carotid Stent (PERFORMANCE 1 Trial)
Brief Title: Evaluation of the 3-in-1 Neuroguard IEP System for Carotid Artery Stenosis
Acronym: PERFORMANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contego Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP1263
Record Dates: First submitted 2019-07-26; First posted 2019-10-29 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid artery stenting with Neuroguard IEP System (Experimental): To evaluate the safety and feasibility of the Neuroguard IEP System when used in patients with clinically significant carotid artery stenosis requiring revascularization.
  Interventions: Device: Neuroguard® IEP 3-in-1 Carotid Stent and Post-Dilation Balloon System with Integrated Embolic Protection (Neuroguard IEP System)

INTERVENTIONS:
Device: Neuroguard® IEP 3-in-1 Carotid Stent and Post-Dilation Balloon System with Integrated Embolic Protection (Neuroguard IEP System) — The Neuroguard® IEP 3-in-1 Carotid Stent and Post-Dilation Balloon System with Integrated Embolic Protection is indicated for improving the carotid luminal diameter in patients with clinically significant carotid artery stenosis and for the simultaneous capture and removal of embolic material during angioplasty and stenting.

SUMMARY:
The Neuroguard IEP System is a 3-in-1 carotid stent delivery system consisting of an angioplasty balloon, an integrated embolic protection device and a nitinol self-expanding stent loaded over the balloon and constrained by an outer sheath. The PERFORMANCE I study is a multi-center, prospective, single arm open label study to evaluate the safety and feasibility of the Neuroguard IEP System for the treatment of carotid artery stenosis. The primary endpoint will be the proportion of patients with Major Adverse Events (MAE) reported within 30 days from the index procedure.

The primary objective of the PERFORMANCE I study is to evaluate the safety and feasibility of the Neuroguard IEP Carotid Stent System when used in patients with clinically significant carotid artery stenosis requiring revascularization.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-breastfeeding female subjects whose age is ≥18 years.
2. Patient is willing and capable of complying with all study protocol requirements, including specified follow-up period and can be contacted by telephone.
3. Patient is willing to provide written informed consent prior to enrollment in study.
4. Females of childbearing potential must have documented negative pregnancy test within 7 days of the Index procedure.
5. Patient is either:

   * Symptomatic with carotid stenosis ≥50% as determined by angiography using NASCET methodology. Symptomatic is defined as transient ischemia attack (TIA) or non-disabling stroke within 180 days of the procedure within the hemisphere supplied by the target vessel; or
   * Asymptomatic with carotid stenosis ≥80% as determined by angiography using NASCET methodology.

7. Patient has a target lesion located at the carotid bifurcation and/or proximal internal carotid artery (ICA).

8. Patient has a single de novo or restenotic (post carotid endarterectomy [CEA]) target lesion or severe tandem lesions close enough that can be covered by a single Neuroguard stent.

9. Target lesion reference vessel diameter between 4.0 and 7.0 mm. 10. Distal vessel diameter at the site of filter deployment between 4.0 mm and 7.0 mm.

11. Sufficient landing zone in the cervical internal carotid artery distal to the lesion to allow for the safe and successful deployment of the primary embolic protection filter (commercially available) and the Neuroguard integrated embolic protection filter.

Exclusion Criteria

1. Life expectancy of less than one year.
2. Patient is experiencing (or has experienced) an evolving, acute, or recent disabling stroke in the last 30 days.
3. Recently (<30 days) implanted heart valve (either surgically or endovascularly) which is a known source of emboli as confirmed on echocardiogram and anticipated or potential cardiovascular sources of emboli that are not adequately treated with anticoagulants .
4. History of or current atrial fibrillation or atrial flutter, including paroxysmal atrial fibrillation.
5. Patient has had an acute myocardial infarction within 72 hours prior to index procedure .
6. Patient has had or has plans to have any major surgical procedure (i.e. intraabdominal or intrathoracic surgery or any surgery/interventional procedure involving cardiac or vascular system) within 30 days before or after the index procedure.
7. Patient has known severe carotid stenosis or complete occlusion contralateral to the target lesion requiring treatment within 30 days following the index procedure.
8. Patient has a modified Rankin Scale (mRS) >2 or has another neurological deficit not due to stroke that may confound the neurological patient assessments (e.g. intracranial tumor).
9. Patient has chronic renal insufficiency (serum creatinine ≥2.5 ml/dL), end stage renal disease on hemodialysis, a history of severe hepatic impairment or malignant hypertension.
10. Patient has platelet count < 100,000/uL.
11. Active bleeding diathesis, hypercoagulable state, or unable to receive blood transfusions.
12. Patient has a history of intolerance or contraindication to standard of care study medications, including antiplatelet therapy.
13. Patient has a known hypersensitivity to nickel or titanium.
14. Sensitivity to heparin or previous incidence of HIT type II.
15. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months, or uncorrected bleeding disorders.
16. Currently enrolled in another interventional device or investigational medication study that has not yet reached the primary endpoint.
17. Patient has a total occlusion of the target carotid artery.
18. Patient has a previously placed stent in the ipsilateral carotid artery.
19. Patient has excessive vascular tortuosity that may preclude the safe introduction of the sheath, guiding catheter, integrated embolic protection device (EPD) or stent.
20. Patient has severe calcification of the target lesion that may prevent full expansion of the carotid stent.
21. Intraluminal mobile filling defect or fresh thrombus in the target lesion.
22. Occlusion or presence of a string sign in the ipsilateral common or internal carotid artery.
23. Carotid (intracranial) stenosis located distal to the target lesion that is more severe than the target lesion.
24. Known mobile plaque or thrombus in the aortic arch.
25. Patient has a type III aortic arch.
26. Arteriovenous malformations of the territory of the target carotid artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Major Adverse Event (MAE) | 30 days
  Death, stroke, myocardial infarction (MI) within 30 days of the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Cremonesi, MD, Principal Investigator — Maria Cecelia Hospital Cotignola
Locations (6):
- Germany (4):
  - Sankt Gertrauden-Krankenhaus GmbH, Berlin
  - Cardiovascular Centre Frankfurt, Frankfurt
  - Medizinisches Versorgungszentrum, Hamburg
  - Universitätsklinikum Leipzig, Leipzig
- Italy (2):
  - Maria Cecelia Hospital, Cotignola
  - Università Frederico II, Naples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langhoff R, Petrov I, Kedev S, Milosevic Z, Schmidt A, Scheinert D, Schofer J, Sievert H, Sedgewick G, Saylors E, Sachar R, Cremonesi A, Micari A. PERFORMANCE 1 study: Novel carotid stent system with integrated post-dilation balloon and embolic protection device. Catheter Cardiovasc Interv. 2022 Nov;100(6):1090-1099. doi: 10.1002/ccd.30410. Epub 2022 Oct 13. PMID 36229946